CLINICAL TRIAL: NCT02628444
Title: Immunogenicity and Safety of Tetravalent Dengue Vaccine Given in 1-, 2-, or 3- Dose Schedules (STAGE I) Followed by a Single Booster Injection of the Same Vaccine (STAGE II) 1 or 2 Years After the Last Primary Dose in Healthy Subjects 9 to 50 Years of Age in Colombia and the Philippines
Brief Title: Immunogenicity and Safety of Different Vaccination Schedules of Tetravalent Dengue Vaccine in Healthy Subjects 9 to 50 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CYD65; U1111-1161-3242 (Other: WHO); 2020-002854-25 (EudraCT Number)
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Results first posted 2021-02-23 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Dengue Fever; Dengue Hemorrhagic Fever
Keywords: Dengue Fever; Dengue virus; Dengue Hemorrhagic Fever; CYD Dengue Vaccine
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- STAGE-I Group 1: CYD Dengue Vaccine (Experimental): Participants received 3 doses of CYD dengue vaccine 0.5 milliliters (mL) subcutaneously (SC) at Day 0 (Vaccination 1), Month 6 (Vaccination 2), and Month 12 (Vaccination 3).
  Interventions: Biological: CYD Dengue Vaccine
- STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12) (Experimental): Participants received a dose of placebo at Day 0 (Vaccination 1) along with 2 doses of CYD dengue vaccine 0.5 mL SC at Month 6 (Vaccination 2) and Month 12 (Vaccination 3).
  Interventions: Biological: CYD Dengue Vaccine; Biological: Placebo (Sodium chloride 0.9%)
- STAGE-I Group 3: Placebo + CYD Dengue Vaccine (Month 12) (Experimental): Participants received 2 doses of placebo at Day 0 (Vaccination 1) and Month 6 (Vaccination 2) along with a dose of CYD dengue vaccine 0.5 mL SC at Month 12 (Vaccination 3).
  Interventions: Biological: CYD Dengue Vaccine; Biological: Placebo (Sodium chloride 0.9%)
- STAGE-II Group 1a: CYD Vaccine + CYD Booster Vaccine (1 Year) (Experimental): Participants from Group 1 who received vaccination in STAGE-I; and were seropositive at Baseline received a booster dose of CYD dengue vaccine in STAGE-II at 1 year post last dose in STAGE-I (i.e., at Month 24).
  Interventions: Biological: CYD Dengue Vaccine
- STAGE-II Group 2a: Placebo + CYD + CYD Booster (1 Year) (Experimental): Participants from Group 2 who received vaccination in STAGE-I and were seropositive at baseline received a booster injection of CYD dengue vaccine in STAGE-II at 1 year post last dose in STAGE-I (i.e., at Month 24).
  Interventions: Biological: CYD Dengue Vaccine; Biological: Placebo (Sodium chloride 0.9%)
- STAGE-II Group 3a: Placebo + CYD + CYD Booster (1 Year) (Experimental): Participants from Group 3 who received vaccination in STAGE-I and were seropositive at Baseline received a booster injection of CYD dengue vaccine in STAGE-II at 1 year post last dose in STAGE-I (i.e., at Month 24).
  Interventions: Biological: CYD Dengue Vaccine; Biological: Placebo (Sodium chloride 0.9%)
- STAGE-II Group 1b: CYD Vaccine + CYD Booster Vaccine (2 Years) (Experimental): Participants from Group 1 who received vaccination in STAGE-I and were seropositive at Baseline received a booster injection of CYD dengue vaccine in STAGE-II at 2 years post last dose in STAGE-I (i.e., at Month 36).
  Interventions: Biological: CYD Dengue Vaccine
- STAGE-II Group 2b: Placebo + CYD + CYD Booster (2 Years) (Experimental): Participants from Group 2 who received vaccination in STAGE-I and were seropositive at Baseline received a booster injection of CYD dengue vaccine in STAGE-II at 2 years post last dose in STAGE-I (i.e., at Month 36).
  Interventions: Biological: CYD Dengue Vaccine; Biological: Placebo (Sodium chloride 0.9%)
- STAGE-II Group 3b: Placebo + CYD + CYD Booster (2 Years) (Experimental): Participants from Group 3 who received vaccination in STAGE-I and were seropositive at baseline received a booster injection of CYD dengue vaccine in STAGE-II at 2 years post last dose in STAGE-I (i.e., at Month 36).
  Interventions: Biological: CYD Dengue Vaccine; Biological: Placebo (Sodium chloride 0.9%)

INTERVENTIONS:
Biological: CYD Dengue Vaccine — 0.5 mL, Subcutaneous
Biological: Placebo (Sodium chloride 0.9%) — 0.5 mL, Subcutaneous
  Arms: STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12); STAGE-I Group 3: Placebo + CYD Dengue Vaccine (Month 12); STAGE-II Group 2a: Placebo + CYD + CYD Booster (1 Year); STAGE-II Group 2b: Placebo + CYD + CYD Booster (2 Years); STAGE-II Group 3a: Placebo + CYD + CYD Booster (1 Year); STAGE-II Group 3b: Placebo + CYD + CYD Booster (2 Years)

SUMMARY:
The aim of the study was to assess the immune response and the safety of different vaccination schedules of CYD dengue vaccine.

The primary objectives of the study were:

* To demonstrate the non-inferiority of the immune response elicited against each dengue serotype by CYD dengue vaccine given as a 2-dose schedule (Group 2) compared to the immune response elicited by CYD dengue vaccine given as a 3-dose schedule (Group 1), in previously dengue exposed participants 28 days after the last injection.
* To demonstrate the non-inferiority of the immune response elicited against each dengue serotype by CYD dengue vaccine given as a 2-dose schedule (Group 2) compared to the immune response elicited by CYD vaccine given as a 3-dose schedule (Group 1) in previously dengue exposed participants, 1 year after the last injection.
* To demonstrate the non-inferiority of the immune response elicited against each dengue serotype elicited by a booster dose of CYD dengue vaccine one year or two years after the last injection in the primary series in previously dengue exposed participants, compared to the immune response post dose 3 in Group 1.

The secondary objectives of the study were:

* To demonstrate the superiority of the immune response elicited by CYD dengue vaccine given as a 2-dose schedule (Group 2) compared to the immune response elicited by CYD dengue vaccine given as a 3-dose schedule (Group 1), in previously dengue exposed participants, 28 days after the last injection.
* To demonstrate the superiority of the immune response elicited by CYD dengue vaccine given as a 2-dose schedule (Group 2) compared to the immune response elicited by CYD dengue vaccine given as a 3-dose schedule (Group 1), in previously dengue exposed participants, one year after the last injection.
* To describe the neutralizing antibody levels of each dengue serotype at 28 days post-injection 3 to the antibody levels immediately before receiving a booster dose, by baseline dengue serostatus.
* To describe the neutralizing antibody levels of each dengue serotype at 28 days post-injection 2 and 28 days post-injection 3 from Group 1 in a primary series schedule by baseline dengue serostatus.
* To demonstrate the superiority of the immune response elicited against each dengue serotype 28 days after administration of a booster dose of CYD dengue vaccine, in previously dengue exposed participants, at one year or two years after last injection in the primary series.
* To describe the seroconversion rate 28 days post-booster injection in all 3 groups.
* To describe all hospitalized virologically confirmed dengue (VCD) cases during the study.
* To evaluate the safety profile of CYD after each and any injection during the trial. Safety assessments include solicited reactions within 7 or 14 days after each injection, unsolicited adverse events within 28 days after each injection, and serious adverse events during the study period.

DETAILED DESCRIPTION:
Healthy participants aged between 9 and 50 year received CYD dengue vaccine in various schedules, in two sequential stages. In the first stage, participants received 1, 2 or 3 injections of CYD dengue vaccine over a 12-month period. In the second stage, participants were randomized to receive a booster dose of CYD dengue vaccine at either 12 months (Subgroup a) or 24 months (Subgroup b) after the third injection of study vaccine. During the conduction of this trial, the World Health Organization (WHO) indication about vaccinating only baseline seropositive participants was arisen; at this moment, STAGE I of the trial was completed. For STAGE II, only participants who were previously dengue exposed at baseline (dengue seropositive) were eligible to receive the booster dose.

ELIGIBILITY:
Inclusion Criteria:

* Aged 9 to 50 years on the day of enrollment.
* Participant in good health, based on medical history and physical examination.
* Assent form or informed consent form (ICF) had been signed and dated by the participant (based on local regulations), and ICF had been signed and dated by the parent(s) or another legally acceptable representative (and by an independent witness if required by local regulations).
* Participant and parent(s)/legally acceptable representative(s) were able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Participant was pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination until at least 4 weeks after the last vaccination).
* Participation at the time of study enrollment (or in the 4 weeks preceding the first trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device or medical procedure.
* Self-reported or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Self-reported systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances.
* Chronic illness that, in the opinion of the investigator, was at a stage where it might interfere with trial conduct or completion.
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response.
* Planned receipt of any vaccine in the 4 weeks following any trial vaccination.
* Previous vaccination against dengue disease with either the trial vaccine or another vaccine.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction that, based on investigator's judgment, might interfere with the participant's ability to comply with trial procedures.
* Identified as a site employee of the Investigator, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members (i.e., immediate, husband, wife, and their children, adopted or natural) of the employees or the Investigator.
* A prospective participant must not be included in the study until the following conditions and/or symptoms were resolved:

  * Febrile illness (temperature greater than or equal to [>=] 38.0 degree Celsius) or moderate or severe acute illness/infection (according to Investigator's judgment) on the day of vaccination.
  * Receipt of any vaccine in the 4 weeks preceding the first trial vaccination.

Ages: 9 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1050 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (6):
- Colombia (3):
  - Investigational Site 102, Barranquilla
  - Investigational Site 101, Cali
  - Investigational Site 103, Medellín
- Philippines (3):
  - Investigational Primary Site Muntinlupa 201_Satellite Site San Pablo 202, City of Muntinlupa
  - Investigational Site 203, Manila
  - Investigational Site 204, Manila

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Coronel-Martinez DL, Park J, Lopez-Medina E, Capeding MR, Bonfanti AAC, Montalban MC, Ramirez I, Gonzales MLA, Zambrano B, Dayan G, Chen Z, Wang H, Bonaparte M, Rojas A, Ramirez JC, Verdan MA, Noriega F. Immunogenicity and safety of booster CYD-TDV dengue vaccine after alternative primary vaccination schedules in healthy individuals aged 9-50 years: a randomised, controlled, phase 2, non-inferiority study. Lancet Infect Dis. 2022 Jun;22(6):901-911. doi: 10.1016/S1473-3099(21)00706-4. Epub 2022 Mar 29. PMID 35364022
- [Derived] Coronel-MartInez DL, Park J, Lopez-Medina E, Capeding MR, Cadena Bonfanti AA, Montalban MC, Ramirez I, Gonzales MLA, DiazGranados CA, Zambrano B, Dayan G, Savarino S, Chen Z, Wang H, Sun S, Bonaparte M, Rojas A, Ramirez JC, Verdan MA, Noriega F. Immunogenicity and safety of simplified vaccination schedules for the CYD-TDV dengue vaccine in healthy individuals aged 9-50 years (CYD65): a randomised, controlled, phase 2, non-inferiority study. Lancet Infect Dis. 2021 Apr;21(4):517-528. doi: 10.1016/S1473-3099(20)30767-2. Epub 2020 Nov 16. PMID 33212067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 active centers in 2 countries. A total of 1050 participants were enrolled from 02 May 2016 to 16 September 2016.
Pre-assignment Details: Participants were enrolled and randomized in 1:1:1 ratio to 1 of 3 treatment arms in STAGE-I. After STAGE-I, participants identified as seropositive at Baseline were randomized in ratio 1:1 to 1 of 2 subgroups (a [1a, 2a, 3a] or b [1b, 2b, 3b]) and received one CYD booster vaccine in STAGE-II at either 12 months (Subgroup a) or 24 months (Subgroup b) post last vaccination in STAGE-I. Here, 'M' in the period titles signifies months.
Groups:
- STAGE-II Group 1a: CYD Vaccine + CYD Booster Vaccine (1 Year): Participants from Group 1 who received vaccination in STAGE-I and were seropositive at Baseline received a booster dose of CYD dengue vaccine in STAGE-II at 1 year post last dose in STAGE-I (i.e., at Month 24).
Period: Stage-I(24M:12M Treatment+12M Follow-up)
Arm/Group | STAGE-I Group 1: CYD Dengue Vaccine | STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12) | STAGE-I Group 3: Placebo + CYD Dengue Vaccine (Month 12) | STAGE-II Group 1a: CYD Vaccine + CYD Booster Vaccine (1 Year) | STAGE-II Group 2a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 3a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 1b: CYD Vaccine + CYD Booster Vaccine (2 Years) | STAGE-II Group 2b: Placebo + CYD + CYD Booster (2 Years) | STAGE-II Group 3b: Placebo + CYD + CYD Booster (2 Years)
Started (Randomized) | 350 | 348 | 352 | 0 | 0 | 0 | 0 | 0 | 0
Vaccinated | 348 | 348 | 352 | 0 | 0 | 0 | 0 | 0 | 0
Full Analysis Set (FAS) (FAS population included participants who had received either at least 1 injection of CYD dengue vaccine or placebo; and had at least 1 blood sample drawn and valid post-vaccination serology results.) | 333 | 328 | 332 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 314 | 309 | 310 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 36 | 39 | 42 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse event (AE) intensity less than (<) Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Serious AE (SAE) | 0 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Voluntary withdrawal not due to AE | 21 | 16 | 25 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance with protocol | 9 | 16 | 9 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 3 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Period: STAGE-II(18M:12M Treatment+6M Follow-up)
Arm/Group | STAGE-I Group 1: CYD Dengue Vaccine | STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12) | STAGE-I Group 3: Placebo + CYD Dengue Vaccine (Month 12) | STAGE-II Group 1a: CYD Vaccine + CYD Booster Vaccine (1 Year) | STAGE-II Group 2a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 3a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 1b: CYD Vaccine + CYD Booster Vaccine (2 Years) | STAGE-II Group 2b: Placebo + CYD + CYD Booster (2 Years) | STAGE-II Group 3b: Placebo + CYD + CYD Booster (2 Years)
Started (Started indicates the number of participants who were enrolled and randomized dengue seropositive subjects at baseline.) | 0 | 0 | 0 | 145 | 152 | 157 | 149 | 152 | 151
Vaccinated | 0 | 0 | 0 | 55 | 59 | 62 | 53 | 56 | 53
Completed | 0 | 0 | 0 | 55 | 59 | 62 | 53 | 54 | 52
Not Completed | 0 | 0 | 0 | 90 | 93 | 95 | 96 | 98 | 99
Not completed — Other AE | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance with protocol | 0 | 0 | 0 | 83 | 83 | 83 | 81 | 84 | 85
Not completed — Voluntary withdrawal not due to AE | 0 | 0 | 0 | 5 | 6 | 10 | 12 | 11 | 9
Not completed — SAE | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized population.
Groups:
- STAGE-I Group 1: CYD Dengue Vaccine: Participants received 3 doses of CYD dengue vaccine 0.5 mL SC at Day 0 (Vaccination 1), Month 6 (Vaccination 2), and Month 12 (Vaccination 3).
- Total: Total of all reporting groups
Arm/Group | STAGE-I Group 1: CYD Dengue Vaccine | STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12) | STAGE-I Group 3: Placebo + CYD Dengue Vaccine (Month 12) | Total
Number analyzed (Participants) | 350 | 348 | 352 | 1050
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (14.42) | 31.3 (14.47) | 31.1 (14.62) | 31.1 (14.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 197 | 185 | 572
  Male | 160 | 151 | 167 | 478
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 171 | 172 | 169 | 512
  Asian | 174 | 172 | 177 | 523
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 6 | 14
  White | 0 | 1 | 0 | 1
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Dengue Baseline Status [Count of Participants; unit: Participants] — Baseline dengue seropositive participants: participants with greater than equal to (>=) 10 (1/dilution) for at least 1 serotype with parental dengue virus strain. Baseline dengue seronegative participants were defined as participants with valid titer less than (<) 10 (1/dilution) for all serotypes with parental dengue virus strains. Baseline dengue status was evaluated in FAS population that included participants who had received either at least 1 injection of either CYD dengue vaccine or placebo and had at least 1 blood sample drawn and valid post-injection serology results.
  Participants
    Seropositive participants | 281 | 288 | 291 | 860
    Seronegative participants | 52 | 40 | 41 | 133
    Undetermined | 17 | 20 | 20 | 57

OUTCOME MEASURES:

1. Primary Outcome: STAGE-I: Geometric Mean Titers (GMTs) Against Each Dengue Virus Serotype 28 Days After Last CYD Dengue Vaccination in Participants Who Were Seropositive at Baseline
Description: GMTs of antibodies against each of the 4 dengue virus serotypes (1, 2, 3, or 4) were assessed using plaque reduction neutralization test (PRNT) assay method. Titers were measured in terms of 1/dilution. Dengue seropositive participants at Baseline was defined as participants with titers >=10 (1/dilution) for at least 1 serotype with parental dengue virus strains. Per-protocol analysis set (PPAS) included all participants who had no protocol violations; and who met any of following study violations were excluded from PPAS (STAGE I/II): had not met all protocol-specified inclusion/exclusion criteria, had not received correct doses or injections, received vaccine other than randomized schedule, did not receive vaccination in proper time window, had not provided post-dose serology sample in proper time window, received protocol-restricted medication, therapy, or vaccine.
Time Frame: 28 days after last CYD dengue vaccination
Population: Analysis performed on PPAS. Here, 'Overall number of participant analyzed'=participants with available data for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for Group 3, as pre-specified in protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | STAGE-I Group 1: CYD Dengue Vaccine | STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12)
Number analyzed (Participants) | 265 | 272
titers
  Serotype 1 | 822 [700 to 964] | 899 [752 to 1075]
  Serotype 2 | 875 [770 to 995] | 869 [754 to 1002]
  Serotype 3 | 610 [535 to 694] | 599 [524 to 685]
  Serotype 4 | 531 [470 to 601] | 510 [453 to 575]
Statistical Analysis 1: Comparison: STAGE-I Group 1: CYD Dengue Vaccine vs STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12); Group 2/Group 1: Serotype 1; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the two-sided 95% confidence interval (CI) of the ratio of GMTs between groups (Group 2/Group 1) was greater than (>) 1/2. Overall non-inferiority was demonstrated if all 4 serotypes achieved non-inferiority; GMT Ratio = 1.09, 95% CI 2-sided [0.862 to 1.39]
Statistical Analysis 2: Comparison: STAGE-I Group 1: CYD Dengue Vaccine vs STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12); Group 2/Group 1: Serotype 2; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the two-sided 95% CI of the ratio of GMTs between groups (Group 2/Group 1) was >1/2. Overall non-inferiority was demonstrated if all 4 serotypes achieved non-inferiority; GMT Ratio = 0.993, 95% CI 2-sided [0.820 to 1.20]
Statistical Analysis 3: Comparison: STAGE-I Group 1: CYD Dengue Vaccine vs STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12); Group 2/Group 1: Serotype 3; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT Ratio = 0.983, 95% CI 2-sided [0.816 to 1.18]
Statistical Analysis 4: Comparison: STAGE-I Group 1: CYD Dengue Vaccine vs STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12); Group 2/Group 1: Serotype 4; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 0.960, 95% CI 2-sided [0.809 to 1.14]

2. Primary Outcome: STAGE-I: Geometric Mean Titers Against Each Dengue Virus Serotype 1 Year After Last CYD Dengue Vaccination in Participants Who Were Seropositive at Baseline
Description: GMTs of antibodies against each of the 4 dengue virus serotypes (1, 2, 3 or 4) were assessed using the PRNT assay method. Titers were measured in terms of 1/dilution. Dengue seropositive participants at Baseline were defined as participants with titers >=10 (1/dilution) for at least one serotype with the parental dengue virus strains.
Time Frame: 1 year after last CYD dengue vaccination
Population: Analysis was performed on PPAS. Here, 'Overall number of participant analyzed'=participants with available data for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for Group 3, as pre-specified in protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | STAGE-I Group 1: CYD Dengue Vaccine | STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12)
Number analyzed (Participants) | 185 | 190
titers
  Serotype 1 | 490 [398 to 604] | 504 [403 to 630]
  Serotype 2 | 821 [704 to 957] | 737 [611 to 888]
  Serotype 3 | 477 [405 to 561] | 437 [368 to 519]
  Serotype 4 | 270 [235 to 310] | 238 [205 to 277]
Statistical Analysis 1: Comparison: STAGE-I Group 1: CYD Dengue Vaccine vs STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12); Group 2/Group 1: Serotype 1; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT Ratio = 1.03, 95% CI 2-sided [0.757 to 1.40]
Statistical Analysis 2: Comparison: STAGE-I Group 1: CYD Dengue Vaccine vs STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12); Group 2/Group 1: Serotype 2; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT Ratio = 0.897, 95% CI 2-sided [0.705 to 1.14]
Statistical Analysis 3: Comparison: STAGE-I Group 1: CYD Dengue Vaccine vs STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12); Group 2/Group 1: Serotype 3; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT Ratio = 0.917, 95% CI 2-sided [0.724 to 1.16]
Statistical Analysis 4: Comparison: STAGE-I Group 1: CYD Dengue Vaccine vs STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12); Group 2/Group 1: Serotype 4; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT Ratio = 0.884, 95% CI 2-sided [0.720 to 1.09]

3. Primary Outcome: STAGE-II: Geometric Mean Titers Against Each Dengue Virus Serotype Within Group 1a and Group 1 After the Third Dose of CYD Dengue Vaccination in Participants Who Were Seropositive at Baseline
Description: GMTs of antibodies against each of the 4 dengue virus serotypes (1, 2, 3 or 4) were assessed using the PRNT assay method. Titers were measured in terms of 1/dilution. Dengue seropositive participants at Baseline were defined as participants with titers >=10 (1/dilution) for at least one serotype with the parental dengue virus strains. Data of Group 1 (28 days post-dose 3 in STAGE-I) and Group 1a (28 days 12 months Booster dose) were reported and compared in this outcome measure. GMT paired ratio (given in statistical analysis section) was calculated by dividing geometric mean values of Group 1a: 28 days post 12 months booster dose in STAGE-II by Group 1: 28 days post-dose 3 in STAGE-I.
Time Frame: Group 1: 28 days post-dose 3 in STAGE-I, Group 1a: 28 days post 12 months booster dose in STAGE-II
Population: Analysis was performed on PPAS. Here, 'Overall number of participant analyzed'=participants with available data for this outcome measure.
Measure: Geometric Mean (98.75% Confidence Interval); unit: titers
Groups:
- Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I: Participants who received 3 doses of CYD dengue vaccine in STAGE-I, and were seropositive at Baseline were assessed 28 days after third CYD vaccine in STAGE-I.
- Group 1a: CYD Dengue Vaccine-28 Days Post 12 Month Booster Dose: Participants from Group 1 (STAGE-I) who were seropositive at Baseline and received a booster dose at 1 year (or 12 months) post last dose in STAGE-I, were assessed 28 days after CYD dengue booster dose vaccination.
Arm/Group | Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I | Group 1a: CYD Dengue Vaccine-28 Days Post 12 Month Booster Dose
Number analyzed (Participants) | 53 | 53
titers
  Serotype 1 | 853 [526 to 1384] | 483 [281 to 832]
  Serotype 2 | 1186 [809 to 1738] | 884 [602 to 1300]
  Serotype 3 | 696 [483 to 1002] | 722 [458 to 1140]
  Serotype 4 | 592 [400 to 876] | 383 [269 to 545]
Statistical Analysis 1: Comparison: Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I vs Group 1a: CYD Dengue Vaccine-28 Days Post 12 Month Booster Dose; Group 1a Booster/Group 1 Post-dose 3: Serotype 1; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the two-sided 95% CI of the ratio of GMTs within groups (Group 1a Booster/Group 1) was >1/2. Overall non-inferiority was demonstrated if all 4 serotypes achieved non-inferiority; GMT paired ratio = 0.567, 98.75% CI 2-sided [0.399 to 0.805]
Statistical Analysis 2: Comparison: Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I vs Group 1a: CYD Dengue Vaccine-28 Days Post 12 Month Booster Dose; Group 1a Booster/Group 1 Post-dose 3: Serotype 2; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; GMT paired ratio = 0.746, 98.75% CI 2-sided [0.550 to 1.01]
Statistical Analysis 3: Comparison: Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I vs Group 1a: CYD Dengue Vaccine-28 Days Post 12 Month Booster Dose; Group 1a Booster/Group 1 Post-dose 3: Serotype 3; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; GMT paired ratio = 1.04, 98.75% CI 2-sided [0.686 to 1.57]
Statistical Analysis 4: Comparison: Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I vs Group 1a: CYD Dengue Vaccine-28 Days Post 12 Month Booster Dose; Group 1a Booster/Group 1 Post-dose 3: Serotype 4; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; GMT paired ratio = 0.647, 98.75% CI 2-sided [0.434 to 0.963]

4. Primary Outcome: STAGE-II: Geometric Mean Titers Against Each Dengue Virus Serotype Comparison Between Group 2a and Group 1 After the Third Dose of CYD Dengue Vaccination in Participants Who Were Seropositive at Baseline
Description: GMTs of antibodies against each of the 4 dengue virus serotypes (1, 2, 3 or 4) were assessed using the PRNT assay method. Titers were measured in terms of 1/dilution. Dengue seropositive participants at Baseline were defined as participants with titers >=10 (1/dilution) for at least one serotype with the parental dengue virus strains. Data of Group 1 (28 days post-dose 3 in STAGE-I) and Group 2a (28 days post 12 months Booster dose) were reported and compared in this outcome measure. GMT ratio (given in statistical analysis section) was calculated by dividing geometric mean values of Group 2a: 28 days post 12 months booster dose in STAGE-II by Group 1: 28 days Post-dose 3 in STAGE-I.
Time Frame: Group 1: 28 days post-dose 3 in STAGE-I, Group 2a: 28 days post 12 months booster dose in STAGE-II
Population: as for outcome 3
Measure: Geometric Mean (98.75% Confidence Interval); unit: titers
Groups:
- Group 2a: CYD Dengue Vaccine-28 Days Post 12 Months Booster Dose: Participants from Group 2 (STAGE-I) who were seropositive at Baseline and received a booster dose at 1 year (or 12 months) post last dose in STAGE-I, were assessed 28 days after CYD dengue booster dose vaccination.
Arm/Group | Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I | Group 2a: CYD Dengue Vaccine-28 Days Post 12 Months Booster Dose
Number analyzed (Participants) | 112 | 58
titers
  Serotype 1 | 875 [614 to 1248] | 549 [331 to 911]
  Serotype 2 | 1023 [771 to 1356] | 828 [569 to 1203]
  Serotype 3 | 568 [433 to 745] | 676 [436 to 1049]
  Serotype 4 | 540 [418 to 697] | 270 [200 to 364]
Statistical Analysis 1: Comparison: Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I vs Group 2a: CYD Dengue Vaccine-28 Days Post 12 Months Booster Dose; Group 2a Booster dose/Group 1 Post-dose 3: Serotype 1; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the two-sided Bonferroni corrected 95% CI for the ratio of GMTs between groups (Group 2a Booster/Group 1) was >1/2. Overall non-inferiority was demonstrated if all 4 serotypes achieved non-inferiority; GMT Ratio = 0.627, 98.75% CI 2-sided [0.342 to 1.15]
Statistical Analysis 2: Comparison: Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I vs Group 2a: CYD Dengue Vaccine-28 Days Post 12 Months Booster Dose; Group 2a Booster/Group 1 Post-dose 3: Serotype 2; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; GMT Ratio = 0.809, 98.75% CI 2-sided [0.505 to 1.30]
Statistical Analysis 3: Comparison: Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I vs Group 2a: CYD Dengue Vaccine-28 Days Post 12 Months Booster Dose; Group 2a Booster/Group 1 Post-dose 3: Serotype 3; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; GMT Ratio = 1.19, 98.75% CI 2-sided [0.732 to 1.94]
Statistical Analysis 4: Comparison: Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I vs Group 2a: CYD Dengue Vaccine-28 Days Post 12 Months Booster Dose; Group 2a Booster/Group 1 Post-dose 3: Serotype 4; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; GMT Ratio = 0.499, 98.75% CI 2-sided [0.331 to 0.754]

5. Primary Outcome: STAGE-II: Geometric Mean Titers Against Each Dengue Virus Serotype Within Group 1b and Group 1 After the Third Dose of CYD Dengue Vaccination in Participants Who Were Seropositive at Baseline
Description: GMTs of antibodies against each of the 4 dengue virus serotypes (1, 2, 3 or 4) were assessed using the PRNT assay method. Titers were measured in terms of 1/dilution. Dengue seropositive participants at Baseline were defined as participants with titers >=10 (1/dilution) for at least one serotype with the parental dengue virus strains. Data of Group 1 (28 days post-dose 3 in STAGE-I) and Group 1b (28 days post 24 months booster dose) were reported and compared in this outcome measure. GMT paired ratio (given in statistical analysis section) was calculated by dividing geometric mean values of Group 1b: 28 days post 24 months booster dose in STAGE-II by Group 1: 28 days Post-dose 3 in STAGE-I.
Time Frame: Group 1: 28 days post-dose 3 in STAGE-I, Group 1b: 28 days post 24 months booster dose in STAGE-II
Population: as for outcome 3
Measure: Geometric Mean (98.75% Confidence Interval); unit: titers
Groups:
- Group 1b: CYD Dengue Vaccine-28 Days Post 24 Month Booster Dose: Participants from Group 1 (STAGE-I) who were seropositive at Baseline and received a booster dose at 2 years (or 24 months) post last dose in STAGE-I, were assessed 28 days after CYD dengue booster dose vaccination.
Arm/Group | Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I | Group 1b: CYD Dengue Vaccine-28 Days Post 24 Month Booster Dose
Number analyzed (Participants) | 48 | 48
titers
  Serotype 1 | 1017 [592 to 1746] | 700 [401 to 1220]
  Serotype 2 | 838 [554 to 1269] | 730 [497 to 1071]
  Serotype 3 | 486 [333 to 708] | 559 [395 to 792]
  Serotype 4 | 556 [400 to 774] | 364 [260 to 510]
Statistical Analysis 1: Comparison: Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I vs Group 1b: CYD Dengue Vaccine-28 Days Post 24 Month Booster Dose; Group 1b Booster/Group 1 Post-dose 3: Serotype 1; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the two-sided 95% CI of the ratio of GMTs within groups (Group 1b booster/Group 1) was >1/2. Overall non-inferiority was demonstrated if all 4 serotypes achieved non-inferiority; GMT paired ratio = 0.688, 98.75% CI 2-sided [0.479 to 0.989]
Statistical Analysis 2: Comparison: Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I vs Group 1b: CYD Dengue Vaccine-28 Days Post 24 Month Booster Dose; Group 1b Booster/Group 1 Post-dose 3: Serotype 2; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; GMT paired ratio = 0.871, 98.75% CI 2-sided [0.673 to 1.13]
Statistical Analysis 3: Comparison: Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I vs Group 1b: CYD Dengue Vaccine-28 Days Post 24 Month Booster Dose; Group 1b Booster/Group 1 Post-dose 3: Serotype 3; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; GMT paired ratio = 1.15, 98.75% CI 2-sided [0.887 to 1.49]
Statistical Analysis 4: Comparison: Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I vs Group 1b: CYD Dengue Vaccine-28 Days Post 24 Month Booster Dose; Group 1b Booster/Group 1 Post-dose 3: Serotype 4; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; GMT paired ratio = 0.655, 98.75% CI 2-sided [0.471 to 0.911]

6. Primary Outcome: STAGE-II: Geometric Mean Titers Against Each Dengue Virus Serotype Comparison Between Group 2b and Group 1 After the Third Dose of CYD Dengue Vaccination in Participants Who Were Seropositive at Baseline
Description: GMTs of antibodies against each of the 4 dengue virus serotypes (1, 2, 3 or 4) were assessed using the PRNT assay method. Titers were measured in terms of 1/dilution. Dengue seropositive participants at Baseline were defined as participants with titers >=10 (1/dilution) for at least one serotype with the parental dengue virus strains. Data of Group 1 (28 days post-dose 3 in STAGE-I) and Group 2b (28 days post 24 months Booster dose) was reported and compared in this outcome measure. GMT ratio (given in statistical analysis section) was calculated by dividing geometric mean values of Group 2b: 28 days post 24 months booster dose in STAGE-II by Group 1: 28 days post-dose 3 in STAGE-I.
Time Frame: Group 1: 28 days post-dose 3 in STAGE-I, Group 2b: 28 days post 24 months Booster dose in STAGE-II
Population: as for outcome 3
Measure: Geometric Mean (98.75% Confidence Interval); unit: titers
Groups:
- Group 2b: CYD Dengue Vaccine-28 Days Post 24 Month Booster Dose: Participants from Group 1 (STAGE-I) who were seropositive at Baseline and received a booster dose at 2 years (or 24 months) post last dose in STAGE-I, were assessed 28 days after CYD dengue booster dose vaccination.
Arm/Group | Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I | Group 2b: CYD Dengue Vaccine-28 Days Post 24 Month Booster Dose
Number analyzed (Participants) | 112 | 50
titers
  Serotype 1 | 875 [614 to 1248] | 778 [429 to 1414]
  Serotype 2 | 1023 [771 to 1356] | 692 [430 to 1116]
  Serotype 3 | 568 [433 to 745] | 517 [365 to 733]
  Serotype 4 | 540 [418 to 697] | 379 [261 to 551]
Statistical Analysis 1: Comparison: Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I vs Group 2b: CYD Dengue Vaccine-28 Days Post 24 Month Booster Dose; Group 2b Booster/Group 1 Post-dose 3: Serotype 1; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the two-sided 95% CI of the ratio of GMTs between groups (Group 2b Booster/Group 1) was >1/2. Overall non-inferiority was demonstrated if all 4 serotypes achieved non-inferiority; GMT ratio = 0.889, 98.75% CI 2-sided [0.462 to 1.71]
Statistical Analysis 2: Comparison: Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I vs Group 2b: CYD Dengue Vaccine-28 Days Post 24 Month Booster Dose; Group 2b Booster/Group 1 Post-dose 3: Serotype 2; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; GMT ratio = 0.677, 98.75% CI 2-sided [0.402 to 1.14]
Statistical Analysis 3: Comparison: Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I vs Group 2b: CYD Dengue Vaccine-28 Days Post 24 Month Booster Dose; Group 2b Booster/Group 1 Post-dose 3: Serotype 3; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; GMT ratio = 0.911, 98.75% CI 2-sided [0.573 to 1.45]
Statistical Analysis 4: Comparison: Group 1: CYD Dengue Vaccine-28 Days Post-dose 3 in STAGE-I vs Group 2b: CYD Dengue Vaccine-28 Days Post 24 Month Booster Dose; Group 2b Booster/Group 1 Post-dose 3: Serotype 4; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; GMT ratio = 0.702, 98.75% CI 2-sided [0.447 to 1.10]

7. Secondary Outcome: STAGE-I: Geometric Mean Titers Against Each Serotype With the Parental Dengue Virus Strains After CYD Dengue Vaccination in Participants Who Were Seropositive at Baseline-Comparison Between Group 1 and Group 2
Description: as for outcome 2
Time Frame: 28 days and 1 year after last CYD dengue vaccination
Population: Analysis was performed on FAS population included participants who had received either at least 1 injection of CYD dengue vaccine or placebo; and had at least 1 blood sample drawn and valid post-injection serology results. Here,'Overall number of participant analyzed'=participants with available data for this outcome measure and 'Number analyzed'=participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | STAGE-I Group 1: CYD Dengue Vaccine | STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12)
Number analyzed (Participants) | 281 | 288
titers
  28 days after last vaccination: Serotype 1: number analyzed (Participants) | 274 | 282
  28 days after last vaccination: Serotype 1 | 834 [713 to 975] | 877 [737 to 1043]
  28 days after last vaccination: Serotype 2: number analyzed (Participants) | 274 | 282
  28 days after last vaccination: Serotype 2 | 879 [775 to 997] | 870 [758 to 1000]
  28 days after last vaccination: Serotype 3: number analyzed (Participants) | 274 | 282
  28 days after last vaccination: Serotype 3 | 620 [545 to 704] | 602 [529 to 686]
  28 days after last vaccination: Serotype 4: number analyzed (Participants) | 274 | 282
  28 days after last vaccination: Serotype 4 | 527 [467 to 595] | 507 [451 to 570]
  1 year after last vaccination: Serotype 1: number analyzed (Participants) | 192 | 197
  1 year after last vaccination: Serotype 1 | 498 [406 to 611] | 512 [411 to 638]
  1 year after last vaccination: Serotype 2: number analyzed (Participants) | 192 | 197
  1 year after last vaccination: Serotype 2 | 815 [702 to 947] | 747 [622 to 897]
  1 year after last vaccination: Serotype 3: number analyzed (Participants) | 192 | 197
  1 year after last vaccination: Serotype 3 | 477 [407 to 558] | 444 [376 to 525]
  1 year after last vaccination: Serotype 4: number analyzed (Participants) | 192 | 197
  1 year after last vaccination: Serotype 4 | 263 [230 to 302] | 241 [208 to 279]
Statistical Analysis 1: Comparison: STAGE-I Group 1: CYD Dengue Vaccine vs STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12); Group2/Group1: Serotype 1 (28 days after last vaccination); Test type: Superiority — The superiority was demonstrated if the lower limit of the two-sided 95% CI was greater than 1 between groups (Group 2/Group 1). Overall superiority of Group 2 to Group 1 was demonstrated if individual serotype null hypotheses were rejected; GMT Ratio = 1.05, 95% CI 2-sided [0.833 to 1.33]
Statistical Analysis 2: Comparison: STAGE-I Group 1: CYD Dengue Vaccine vs STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12); Group2/Group1: Serotype 2 (28 days after last vaccination); Test type: Superiority — [test comment as in outcome 7, analysis 1]; GMT Ratio = 0.99, 95% CI 2-sided [0.821 to 1.19]
Statistical Analysis 3: Comparison: STAGE-I Group 1: CYD Dengue Vaccine vs STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12); Group2/Group1: Serotype 3 (28 days after last vaccination); Test type: Superiority — [test comment as in outcome 7, analysis 1]; GMT Ratio = 0.972, 95% CI 2-sided [0.810 to 1.17]
Statistical Analysis 4: Comparison: STAGE-I Group 1: CYD Dengue Vaccine vs STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12); Group2/Group1: Serotype 4 (28 days after last vaccination); Test type: Superiority — [test comment as in outcome 7, analysis 1]; GMT Ratio = 0.963, 95% CI 2-sided [0.814 to 1.14]
Statistical Analysis 5: Comparison: STAGE-I Group 1: CYD Dengue Vaccine vs STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12); Group2/Group1: Serotype 1 (1 year after last vaccination); Test type: Superiority — [test comment as in outcome 7, analysis 1]; GMT Ratio = 1.03, 95% CI 2-sided [0.762 to 1.39]
Statistical Analysis 6: Comparison: STAGE-I Group 1: CYD Dengue Vaccine vs STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12); Group2/Group1: Serotype 2 (1 year after last vaccination); Test type: Superiority — [test comment as in outcome 7, analysis 1]; GMT Ratio = 0.917, 95% CI 2-sided [0.724 to 1.16]
Statistical Analysis 7: Comparison: STAGE-I Group 1: CYD Dengue Vaccine vs STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12); Group2/Group1: Serotype 3 (1 year after last vaccination); Test type: Superiority — [test comment as in outcome 7, analysis 1]; GMT Ratio = 0.933, 95% CI 2-sided [0.742 to 1.17]
Statistical Analysis 8: Comparison: STAGE-I Group 1: CYD Dengue Vaccine vs STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12); Group2/Group1: Serotype 4 (1 year after last vaccination); Test type: Superiority — [test comment as in outcome 7, analysis 1]; GMT Ratio = 0.916, 95% CI 2-sided [0.750 to 1.12]

8. Secondary Outcome: STAGE-I: Geometric Mean Titers Against Each Serotype With the Parental Dengue Virus Strains in All Participants
Description: GMTs of antibodies against each of the 4 dengue virus serotypes (parental strains) were assessed using the PRNT assay method.
Time Frame: Baseline, 28 days post vaccination 3, and 1 year post vaccination 3
Population: Analysis was performed on FAS. Here, 'Number analyzed'=participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | STAGE-I Group 1: CYD Dengue Vaccine | STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12) | STAGE-I Group 3: Placebo + CYD Dengue Vaccine (Month 12)
Number analyzed (Participants) | 333 | 328 | 332
titers
  Serotype 1: Baseline | 131 [103 to 165] | 187 [147 to 237] | 198 [157 to 250]
  Serotype 1: 28 days post vaccination 3: number analyzed (Participants) | 326 | 322 | 324
  Serotype 1: 28 days post vaccination 3 | 497 [410 to 602] | 586 [482 to 714] | 735 [589 to 916]
  Serotype 1: 1 year post vaccination 3: number analyzed (Participants) | 231 | 232 | 230
  Serotype 1: 1 year post vaccination 3 | 259 [200 to 336] | 279 [213 to 365] | 331 [252 to 435]
  Serotype 2: Baseline | 172 [138 to 214] | 202 [163 to 252] | 181 [147 to 222]
  Serotype 2: 28 days post vaccination 3: number analyzed (Participants) | 326 | 322 | 324
  Serotype 2: 28 days post vaccination 3 | 567 [482 to 666] | 628 [532 to 741] | 734 [614 to 878]
  Serotype 2: 1 year post vaccination 3: number analyzed (Participants) | 231 | 232 | 230
  Serotype 2: 1 year post vaccination 3 | 470 [380 to 582] | 457 [364 to 574] | 500 [402 to 623]
  Serotype 3: Baseline | 163 [131 to 202] | 180 [145 to 222] | 169 [138 to 207]
  Serotype 3: 28 days post vaccination 3: number analyzed (Participants) | 326 | 322 | 324
  Serotype 3: 28 days post vaccination 3 | 432 [373 to 500] | 446 [383 to 519] | 505 [428 to 595]
  Serotype 3: 1 year post vaccination 3: number analyzed (Participants) | 231 | 232 | 230
  Serotype 3: 1 year post vaccination 3 | 294 [240 to 361] | 288 [235 to 354] | 258 [213 to 312]
  Serotype 4: Baseline | 86.7 [71.4 to 105] | 83.8 [69.9 to 100] | 81.2 [67.7 to 97.4]
  Serotype 4: 28 days post vaccination 3: number analyzed (Participants) | 326 | 322 | 324
  Serotype 4: 28 days post vaccination 3 | 429 [380 to 484] | 441 [392 to 496] | 546 [475 to 629]
  Serotype 4: 1 year post vaccination 3: number analyzed (Participants) | 231 | 232 | 230
  Serotype 4: 1 year post vaccination 3 | 203 [176 to 235] | 192 [164 to 226] | 177 [150 to 210]

9. Secondary Outcome: STAGE-I: Geometric Mean Titers Against Each Serotype With the Parental Dengue Virus Strains (by Baseline Dengue Status) in Participants Who Were Seropositive and Seronegative at Baseline
Description: GMTs of antibodies against each of the 4 dengue virus serotypes (1, 2, 3, or 4) were assessed using the PRNT assay method. Titers were measured in terms of 1/dilution. Dengue seropositive participants at Baseline were defined as participants with titers >=10 (1/dilution) for at least one serotype with the parental dengue virus strains. Dengue seronegative participants at Baseline were defined as the participants with valid titer <0 (1/dilution) for all serotypes with parental dengue virus strains.
Time Frame: Baseline, 28 days post vaccination 3, and 1 year post vaccination 3
Population: Analysis was performed on FAS. Here, 'Overall number of participants analyzed'=participants evaluable for this outcome measure and 'Number analyzed'=participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | STAGE-I Group 1: CYD Dengue Vaccine | STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12) | STAGE-I Group 3: Placebo + CYD Dengue Vaccine (Month 12)
Number analyzed (Participants) | 281 | 288 | 291
titers
  Seropositive- Serotype 1: Baseline | 239 [194 to 295] | 304 [244 to 379] | 328 [267 to 404]
  Seropositive- Serotype 1: 28 days post vaccination 3: number analyzed (Participants) | 274 | 282 | 285
  Seropositive- Serotype 1: 28 days post vaccination 3 | 834 [713 to 975] | 877 [737 to 1043] | 1201 [1007 to 1431]
  Seropositive- Serotype 1: 1 year post vaccination 3: number analyzed (Participants) | 192 | 197 | 197
  Seropositive- Serotype 1: 1 year post vaccination 3 | 498 [406 to 611] | 512 [411 to 638] | 618 [500 to 764]
  Seropositive- Serotype 2: Baseline | 331 [279 to 394] | 326 [271 to 393] | 293 [247 to 347]
  Seropositive- Serotype 2: 28 days post vaccination 3: number analyzed (Participants) | 274 | 282 | 285
  Seropositive- Serotype 2: 28 days post vaccination 3 | 879 [775 to 997] | 870 [758 to 1000] | 1046 [912 to 1201]
  Seropositive- Serotype 2: 1 year post vaccination 3: number analyzed (Participants) | 192 | 197 | 197
  Seropositive- Serotype 2: 1 year post vaccination 3 | 815 [702 to 947] | 747 [622 to 897] | 798 [676 to 942]
  Seropositive- Serotype 3: Baseline | 310 [263 to 367] | 290 [241 to 349] | 269 [227 to 319]
  Seropositive- Serotype 3: 28 days post vaccination 3: number analyzed (Participants) | 274 | 282 | 285
  Seropositive- Serotype 3: 28 days post vaccination 3 | 620 [545 to 704] | 602 [529 to 686] | 694 [604 to 797]
  Seropositive- Serotype 3: 1 year post vaccination 3: number analyzed (Participants) | 192 | 197 | 197
  Seropositive- Serotype 3: 1 year post vaccination 3 | 477 [407 to 558] | 444 [376 to 525] | 390 [338 to 450]
  Seropositive- Serotype 4: Baseline | 147 [124 to 174] | 123 [104 to 144] | 118 [100 to 140]
  Seropositive- Serotype 4: 28 days post vaccination 3: number analyzed (Participants) | 274 | 282 | 285
  Seropositive- Serotype 4: 28 days post vaccination 3 | 527 [467 to 595] | 507 [451 to 570] | 581 [507 to 666]
  Seropositive- Serotype 4: 1 year post vaccination 3: number analyzed (Participants) | 192 | 197 | 197
  Seropositive- Serotype 4: 1 year post vaccination 3 | 263 [230 to 302] | 241 [208 to 279] | 227 [194 to 265]
  Seronegative- Serotype 1: Baseline: number analyzed (Participants) | 52 | 40 | 41
  Seronegative- Serotype 1: Baseline | 5.00 [NA to NA] — The 95% CI was not computable as the standard deviation of the sample was 0, since all participants had the same value. | 5.57 [4.65 to 6.67] | 5.49 [4.75 to 6.34]
  Seronegative- Serotype 1: 28 days post vaccination 3: number analyzed (Participants) | 52 | 40 | 39
  Seronegative- Serotype 1: 28 days post vaccination 3 | 32.4 [23.1 to 45.6] | 34.3 [23.8 to 49.4] | 20.2 [12.0 to 34.1]
  Seronegative- Serotype 1: 1 year post vaccination 3: number analyzed (Participants) | 39 | 35 | 33
  Seronegative- Serotype 1: 1 year post vaccination 3 | 10.4 [7.12 to 15.1] | 9.01 [6.30 to 12.9] | 8.04 [5.86 to 11.0]
  Seronegative- Serotype 2: Baseline: number analyzed (Participants) | 52 | 40 | 41
  Seronegative- Serotype 2: Baseline | 5.00 [NA to NA] — The 95% CI was not computable as the standard deviation of the sample was 0, since all participants had the same value. | 6.47 [4.43 to 9.45] | 5.86 [4.99 to 6.89]
  Seronegative- Serotype 2: 28 days post vaccination 3: number analyzed (Participants) | 52 | 40 | 39
  Seronegative- Serotype 2: 28 days post vaccination 3 | 56.2 [40.1 to 78.7] | 63.0 [37.5 to 106] | 55.2 [27.8 to 110]
  Seronegative- Serotype 2: 1 year post vaccination 3: number analyzed (Participants) | 39 | 35 | 33
  Seronegative- Serotype 2: 1 year post vaccination 3 | 31.3 [20.2 to 48.6] | 28.7 [17.3 to 47.7] | 30.9 [17.5 to 54.5]
  Seronegative- Serotype 3: Baseline: number analyzed (Participants) | 52 | 40 | 41
  Seronegative- Serotype 3: Baseline | 5.00 [NA to NA] — The 95% CI was not computable as the standard deviation of the sample was 0, since all participants had the same value. | 5.69 [4.86 to 6.66] | 6.09 [5.05 to 7.34]
  Seronegative- Serotype 3: 28 days post vaccination 3: number analyzed (Participants) | 52 | 40 | 39
  Seronegative- Serotype 3: 28 days post vaccination 3 | 64.2 [48.6 to 84.9] | 53.7 [36.1 to 80.0] | 49.5 [30.1 to 81.5]
  Seronegative- Serotype 3: 1 year post injection 3: number analyzed (Participants) | 39 | 35 | 33
  Seronegative- Serotype 3: 1 year post injection 3 | 27.5 [17.4 to 43.5] | 25.3 [15.8 to 40.3] | 21.8 [13.6 to 35.0]
  Seronegative- Serotype 4: Baseline: number analyzed (Participants) | 52 | 40 | 41
  Seronegative- Serotype 4: Baseline | 5.00 [NA to NA] — The 95% CI was not computable as the standard deviation of the sample was 0, since all participants had the same value. | 5.41 [4.61 to 6.35] | 5.64 [4.90 to 6.50]
  Seronegative- Serotype 4: 28 days post vaccination 3: number analyzed (Participants) | 52 | 40 | 39
  Seronegative- Serotype 4: 28 days post vaccination 3 | 145 [112 to 187] | 164 [114 to 237] | 349 [189 to 646]
  Seronegative- Serotype 4: 1 year post vaccination 3: number analyzed (Participants) | 39 | 35 | 33
  Seronegative- Serotype 4: 1 year post vaccination 3 | 57.1 [42.5 to 76.8] | 53.8 [32.0 to 90.5] | 40.8 [24.9 to 66.8]

10. Secondary Outcome: STAGE-II: Geometric Mean Titers Against Each Serotype With the Parental Dengue Virus Strains After Booster CYD Dengue Vaccination in Participants Seropositive at Baseline
Description: GMTs of antibodies against each of the 4 dengue virus serotype (1, 2, 3, or 4) were assessed using the PRNT assay. Dengue seropositive participants at Baseline were defined as participants with titers >=10 (1/dilution) for at least one serotype with the parental dengue virus strains. Titers were measured in terms of 1/dilution.
Time Frame: Baseline, 28 days post vaccination-3, and 28 days post booster dose
Population: Analysis was performed on FAS. Here, 'Overall number of participant analyzed'=participants with available data for this outcome measure and 'Number analyzed'=participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | STAGE-II Group 1a: CYD Vaccine + CYD Booster Vaccine (1 Year) | STAGE-II Group 2a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 3a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 1b: CYD Vaccine + CYD Booster Vaccine (2 Years) | STAGE-II Group 2b: Placebo + CYD + CYD Booster (2 Years) | STAGE-II Group 3b: Placebo + CYD + CYD Booster (2 Years)
Number analyzed (Participants) | 141 | 144 | 147 | 140 | 144 | 144
titers
  Serotype 1: Baseline | 246 [183 to 331] | 283 [207 to 385] | 309 [227 to 421] | 231 [171 to 313] | 327 [239 to 447] | 350 [265 to 462]
  Serotype 1: 28 days post vaccination 3: number analyzed (Participants) | 137 | 140 | 145 | 137 | 142 | 140
  Serotype 1: 28 days post vaccination 3 | 828 [671 to 1022] | 933 [730 to 1192] | 1111 [868 to 1423] | 840 [664 to 1061] | 824 [644 to 1056] | 1301 [1011 to 1675]
  Serotype 1 : 28 days post booster dose: number analyzed (Participants) | 55 | 59 | 62 | 53 | 54 | 52
  Serotype 1 : 28 days post booster dose | 505 [335 to 763] | 552 [375 to 812] | 861 [572 to 1297] | 707 [472 to 1057] | 749 [465 to 1207] | 1199 [755 to 1902]
  Serotype 2 : Baseline | 370 [295 to 466] | 335 [258 to 437] | 283 [221 to 363] | 296 [228 to 385] | 318 [244 to 413] | 303 [241 to 382]
  Serotype 2 : 28 days post vaccination 3: number analyzed (Participants) | 137 | 140 | 145 | 137 | 142 | 140
  Serotype 2 : 28 days post vaccination 3 | 986 [834 to 1166] | 897 [735 to 1096] | 1018 [850 to 1218] | 783 [648 to 947] | 844 [695 to 1025] | 1077 [871 to 1331]
  Serotype 2 : 28 days post booster dose: number analyzed (Participants) | 55 | 59 | 62 | 53 | 54 | 52
  Serotype 2 : 28 days post booster dose | 856 [638 to 1147] | 858 [639 to 1152] | 867 [640 to 1174] | 813 [600 to 1100] | 655 [461 to 931] | 967 [697 to 1343]
  Serotype 3 : Baseline | 363 [285 to 462] | 399 [308 to 519] | 287 [222 to 371] | 266 [211 to 335] | 210 [164 to 271] | 253 [201 to 317]
  Serotype 3: 28 days post vaccination 3: number analyzed (Participants) | 137 | 140 | 145 | 137 | 142 | 140
  Serotype 3: 28 days post vaccination 3 | 733 [617 to 871] | 659 [547 to 794] | 725 [607 to 865] | 524 [434 to 631] | 551 [459 to 661] | 663 [534 to 823]
  Serotype 3:28 days post booster dose: number analyzed (Participants) | 55 | 59 | 62 | 53 | 54 | 52
  Serotype 3:28 days post booster dose | 721 [511 to 1018] | 667 [477 to 933] | 743 [557 to 992] | 586 [455 to 754] | 477 [364 to 626] | 506 [370 to 691]
  Serotype 4: Baseline | 147 [114 to 190] | 142 [113 to 178] | 115 [89.6 to 146] | 147 [117 to 183] | 106 [84.5 to 133] | 122 [97.3 to 153]
  Serotype 4:28 day post vaccination 3: number analyzed (Participants) | 137 | 140 | 145 | 137 | 142 | 140
  Serotype 4:28 day post vaccination 3 | 512 [433 to 605] | 536 [456 to 631] | 570 [463 to 701] | 543 [456 to 647] | 480 [406 to 568] | 593 [495 to 711]
  Serotype 4 : 28 days post booster dose: number analyzed (Participants) | 55 | 59 | 62 | 53 | 54 | 52
  Serotype 4 : 28 days post booster dose | 380 [292 to 495] | 265 [210 to 334] | 300 [223 to 405] | 368 [290 to 466] | 360 [273 to 474] | 413 [297 to 574]

11. Secondary Outcome: STAGE-I: Percentage of Participants With Antibodies Titer >=10 (1/Dilution) Against Each Serotype With the Parental Dengue Virus Strains in All Participants
Description: GMTs of antibodies against each of the 4 dengue virus serotypes (1, 2, 3 or 4) were assessed using the PRNT assay.
Time Frame: Baseline, 28 days post vaccination 3, and 1 year post vaccination 3
Population: Analysis was performed on FAS. Here, 'Number analyzed'=participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | STAGE-I Group 1: CYD Dengue Vaccine | STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12) | STAGE-I Group 3: Placebo + CYD Dengue Vaccine (Month 12)
Number analyzed (Participants) | 333 | 328 | 332
percentage of participants
  Serotype 1: Baseline | 77.8 [72.9 to 82.1] | 80.5 [75.8 to 84.6] | 83.4 [79.0 to 87.3]
  Serotype 1: 28 days post vaccination 3: number analyzed (Participants) | 326 | 322 | 324
  Serotype 1: 28 days post vaccination 3 | 96.3 [93.7 to 98.1] | 97.2 [94.8 to 98.7] | 94.1 [91.0 to 96.4]
  Serotype 1: 1 year post vaccination 3: number analyzed (Participants) | 231 | 232 | 230
  Serotype 1: 1 year post vaccination 3 | 88.3 [83.5 to 92.2] | 87.5 [82.5 to 91.5] | 88.3 [83.4 to 92.1]
  Serotype 2: Baseline | 82.6 [78.1 to 86.5] | 83.8 [79.4 to 87.7] | 85.2 [81.0 to 88.9]
  Serotype 2: 28 days post vaccination 3: number analyzed (Participants) | 326 | 322 | 324
  Serotype 2: 28 days post vaccination 3 | 98.2 [96.0 to 99.3] | 96.6 [94.0 to 98.3] | 96.0 [93.2 to 97.8]
  Serotype 2: 1 year post vaccination 3: number analyzed (Participants) | 231 | 232 | 230
  Serotype 2: 1 year post vaccination 3 | 95.7 [92.2 to 97.9] | 94.4 [90.6 to 97.0] | 94.8 [91.1 to 97.3]
  Serotype 3: Baseline | 82.6 [78.1 to 86.5] | 84.1 [79.7 to 87.9] | 87.0 [83.0 to 90.5]
  Serotype 3: 28 days post vaccination 3: number analyzed (Participants) | 326 | 322 | 324
  Serotype 3: 28 days post vaccination 3 | 98.5 [96.5 to 99.5] | 98.1 [96.0 to 99.3] | 97.5 [95.2 to 98.9]
  Serotype 3: 1 year post vaccination 3: number analyzed (Participants) | 231 | 232 | 230
  Serotype 3: 1 year post vaccination 3 | 95.7 [92.2 to 97.9] | 95.7 [92.2 to 97.9] | 94.3 [90.5 to 97.0]
  Serotype 4: Baseline | 79.6 [74.8 to 83.8] | 81.4 [76.8 to 85.5] | 81.6 [77.0 to 85.6]
  Serotype 4: 28 days post vaccination 3: number analyzed (Participants) | 326 | 322 | 324
  Serotype 4: 28 days post vaccination 3 | 99.7 [98.3 to 100.0] | 99.4 [97.8 to 99.9] | 98.8 [96.9 to 99.7]
  Serotype 4: 1 year post vaccination 3: number analyzed (Participants) | 231 | 232 | 230
  Serotype 4: 1 year post vaccination 3 | 99.1 [96.9 to 99.9] | 96.6 [93.3 to 98.5] | 95.7 [92.1 to 97.9]

12. Secondary Outcome: STAGE-II: Percentage of Participants With Antibodies Titer >=10 (1/Dilution) Against Each Serotype With the Parental Dengue Virus Strain in Participants Seropositive at Baseline
Description: GMTs of antibodies against each of the 4 dengue virus serotypes (1, 2, 3 or 4) were assessed using the PRNT assay method. Dengue seropositive participants at Baseline were defined as participants with titers >=10 (1/dilution) for at least one serotype with the parental dengue virus strains.
Time Frame: Baseline, 28 days post vaccination 3, and 1 year post vaccination 3
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | STAGE-II Group 1a: CYD Vaccine + CYD Booster Vaccine (1 Year) | STAGE-II Group 2a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 3a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 1b: CYD Vaccine + CYD Booster Vaccine (2 Years) | STAGE-II Group 2b: Placebo + CYD + CYD Booster (2 Years) | STAGE-II Group 3b: Placebo + CYD + CYD Booster (2 Years)
Number analyzed (Participants) | 141 | 144 | 147 | 140 | 144 | 144
percentage of participants
  Serotype 1: Baseline | 92.2 [86.5 to 96.0] | 90.3 [84.2 to 94.6] | 91.8 [86.2 to 95.7] | 92.1 [86.4 to 96.0] | 91.7 [85.9 to 95.6] | 97.2 [93.0 to 99.2]
  Serotype 1: 28 days post vaccination 3: number analyzed (Participants) | 137 | 140 | 145 | 137 | 142 | 140
  Serotype 1: 28 days post vaccination 3 | 100.0 [97.3 to 100.0] | 99.3 [96.1 to 100.0] | 100.0 [97.5 to 100.0] | 99.3 [96.0 to 100.0] | 99.3 [96.1 to 100.0] | 100.0 [97.4 to 100.0]
  Serotype 1 : 1 year post vaccination 3: number analyzed (Participants) | 137 | 138 | 143 | 128 | 130 | 131
  Serotype 1 : 1 year post vaccination 3 | 100.0 [97.3 to 100.0] | 99.3 [96.0 to 100.0] | 99.3 [96.2 to 100.0] | 100.0 [97.2 to 100.0] | 96.9 [92.3 to 99.2] | 98.5 [94.6 to 99.8]
  Serotype 2: Baseline | 99.3 [96.1 to 100.0] | 94.4 [89.3 to 97.6] | 94.6 [89.6 to 97.6] | 96.4 [91.9 to 98.8] | 94.4 [89.3 to 97.6] | 97.2 [93.0 to 99.2]
  Serotype 2 : 28 days post vaccination 3: number analyzed (Participants) | 137 | 140 | 145 | 137 | 142 | 140
  Serotype 2 : 28 days post vaccination 3 | 100.0 [97.3 to 100.0] | 99.3 [96.1 to 100.0] | 100.0 [97.5 to 100.0] | 100.0 [97.3 to 100.0] | 99.3 [96.1 to 100.0] | 100.0 [97.4 to 100.0]
  Serotype 2 : 1 year post vaccination 3: number analyzed (Participants) | 137 | 138 | 143 | 128 | 130 | 131
  Serotype 2 : 1 year post vaccination 3 | 100.0 [97.3 to 100.0] | 99.3 [96.0 to 100.0] | 100.0 [97.5 to 100.0] | 100.0 [97.2 to 100.0] | 98.5 [94.6 to 99.8] | 100.0 [97.2 to 100.0]
  Serotype 3: Baseline | 98.6 [95.0 to 99.8] | 96.5 [92.1 to 98.9] | 95.2 [90.4 to 98.1] | 97.1 [92.8 to 99.2] | 93.1 [87.6 to 96.6] | 100.0 [97.5 to 100.0]
  Serotype 3: 28 days post vaccination: number analyzed (Participants) | 137 | 140 | 145 | 137 | 142 | 140
  Serotype 3: 28 days post vaccination | 100.0 [97.3 to 100.0] | 100.0 [97.4 to 100.0] | 100.0 [97.5 to 100.0] | 99.3 [96.0 to 100.0] | 100.0 [97.4 to 100.0] | 100.0 [97.4 to 100.0]
  Serotype 3 : 1 year post vaccination 3: number analyzed (Participants) | 137 | 138 | 143 | 128 | 130 | 131
  Serotype 3 : 1 year post vaccination 3 | 100.0 [97.3 to 100.0] | 99.3 [96.0 to 100.0] | 99.3 [96.2 to 100.0] | 100.0 [97.2 to 100.0] | 100.0 [97.2 to 100.0] | 100.0 [97.2 to 100.0]
  Serotype 4: Baseline | 93.6 [88.2 to 97.0] | 93.1 [87.6 to 96.6] | 89.8 [83.7 to 94.2] | 95.0 [90.0 to 98.0] | 91.7 [85.9 to 95.6] | 94.4 [89.3 to 97.6]
  Serotype 4: 28 days post vaccination 3: number analyzed (Participants) | 137 | 140 | 145 | 137 | 142 | 140
  Serotype 4: 28 days post vaccination 3 | 100.0 [97.3 to 100.0] | 100.0 [97.4 to 100.0] | 100.0 [97.5 to 100.0] | 100.0 [97.3 to 100.0] | 100.0 [97.4 to 100.0] | 100.0 [97.4 to 100.0]
  Serotype 4: 1 year post vaccination 3: number analyzed (Participants) | 137 | 138 | 143 | 128 | 130 | 131
  Serotype 4: 1 year post vaccination 3 | 100.0 [97.3 to 100.0] | 99.3 [96.0 to 100.0] | 98.6 [95.0 to 99.8] | 100.0 [97.2 to 100.0] | 98.5 [94.6 to 99.8] | 100.0 [97.2 to 100.0]

13. Secondary Outcome: STAGE-I: Number of Participants With Immediate Unsolicited Adverse Events Following Vaccination With CYD Dengue Vaccine or Placebo (Post Any Vaccination)
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the electronic case report form (eCRF) in terms of diagnosis and/or onset post-vaccination. Immediate unsolicited AE were AEs that occurred within 30 minutes after any vaccination.
Time Frame: Within 30 minutes after any vaccination (1, 2, or 3)
Population: Analysis was performed on safety analysis set (SafAS) that included participants who had received at least one injection of either CYD dengue vaccine or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | STAGE-I Group 1: CYD Dengue Vaccine | STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12) | STAGE-I Group 3: Placebo + CYD Dengue Vaccine (Month 12)
Number analyzed (Participants) | 348 | 348 | 352
Participants | 0 | 3 | 0

14. Secondary Outcome: STAGE-II: Number of Participants With Immediate Unsolicited Adverse Events Following Booster Vaccination With CYD Dengue Vaccine
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the eCRF in terms of diagnosis and / or onset post-vaccination. Immediate unsolicited AE were AEs that occurred within 30 minutes after vaccination.
Time Frame: Within 30 minutes after CYD booster vaccination
Population: Analysis was performed on SafAS.
Measure: Count of Participants; unit: Participants
Arm/Group | STAGE-II Group 1a: CYD Vaccine + CYD Booster Vaccine (1 Year) | STAGE-II Group 2a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 3a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 1b: CYD Vaccine + CYD Booster Vaccine (2 Years) | STAGE-II Group 2b: Placebo + CYD + CYD Booster (2 Years) | STAGE-II Group 3b: Placebo + CYD + CYD Booster (2 Years)
Number analyzed (Participants) | 55 | 59 | 62 | 53 | 56 | 53
Participants | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: STAGE-I: Number of Participants With Solicited Injection Site Reactions Following Vaccination With CYD Dengue Vaccine or Placebo (Post Any Vaccination)
Description: Adverse reaction (AR) was defined as all noxious and unintended responses to a medicinal product related to any dose. A Solicited Reaction (SR) was defined as an AR observed and reported under the conditions (symptom and onset) prelisted (i.e., solicited) in the eCRF and considered as related to vaccination. Solicited injection site reaction was an AR at and around the injection site that included pain, erythema, and swelling.
Time Frame: Within 7 days after any vaccination (1, 2, or 3)
Population: Analysis was performed on SafAS. Here, 'Number analyzed'=participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | STAGE-I Group 1: CYD Dengue Vaccine | STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12) | STAGE-I Group 3: Placebo + CYD Dengue Vaccine (Month 12)
Number analyzed (Participants) | 347 | 347 | 352
Participants
  Pain | 109 | 114 | 97
  Erythema | 4 | 3 | 3
  Swelling | 2 | 5 | 5

16. Secondary Outcome: STAGE-I: Number of Participants With Solicited Injection Site Reactions Following Vaccination With CYD Dengue Vaccine or Placebo (Post Each Vaccination)
Description: AR was defined as all noxious and unintended responses to a medicinal product related to any dose. An SR was defined as an AR observed and reported under the conditions (symptom and onset) prelisted (i.e., solicited) in the eCRF and considered as related to vaccination. Solicited injection site reaction was an AR at and around the injection site that included pain, erythema, and swelling.
Time Frame: Within 7 days after each vaccination (1, 2, and 3)
Population: Analysis was performed on SafAS. Here, 'Number analyzed'=participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | STAGE-I Group 1: CYD Dengue Vaccine | STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12) | STAGE-I Group 3: Placebo + CYD Dengue Vaccine (Month 12)
Number analyzed (Participants) | 347 | 347 | 352
Participants
  Post-vaccination 1: Pain | 61 | 61 | 61
  Post-vaccination 1: Erythema | 3 | 3 | 2
  Post vaccination 1: Swelling | 0 | 2 | 2
  Post-vaccination 2: Pain: number analyzed (Participants) | 332 | 328 | 332
  Post-vaccination 2: Pain | 50 | 53 | 50
  Post-vaccination 2: Erythema: number analyzed (Participants) | 332 | 328 | 332
  Post-vaccination 2: Erythema | 1 | 0 | 1
  Post-vaccination 2: Swelling: number analyzed (Participants) | 332 | 328 | 332
  Post-vaccination 2: Swelling | 1 | 1 | 2
  Post-vaccination 3: Pain: number analyzed (Participants) | 325 | 321 | 324
  Post-vaccination 3: Pain | 43 | 49 | 35
  Post-vaccination 3: Erythema: number analyzed (Participants) | 325 | 321 | 324
  Post-vaccination 3: Erythema | 0 | 0 | 1
  Post-vaccination 3: Swelling: number analyzed (Participants) | 325 | 321 | 324
  Post-vaccination 3: Swelling | 1 | 2 | 2

17. Secondary Outcome: STAGE-I: Number of Participants With Solicited Systemic Reactions Following Vaccination With CYD Dengue Vaccine or Placebo (Post Any Vaccination)
Description: An AR was defined as all noxious and unintended responses to a medicinal product related to any dose. An SR was defined as an AR observed and reported under the conditions (symptom and onset) prelisted (i.e., solicited) in the eCRF and considered as related to vaccination. Systemic AEs were all AEs that were not injection site reactions. Solicited systemic reactions included fever, headache, malaise, myalgia, and asthenia.
Time Frame: Within 14 days after any vaccination (1, 2, or 3)
Population: Analysis was performed on SafAS. Here, 'Number analyzed'=participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | STAGE-I Group 1: CYD Dengue Vaccine | STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12) | STAGE-I Group 3: Placebo + CYD Dengue Vaccine (Month 12)
Number analyzed (Participants) | 347 | 347 | 352
Participants
  Fever | 29 | 21 | 31
  Headache | 129 | 122 | 124
  Malaise | 114 | 98 | 102
  Myalgia | 110 | 92 | 86
  Asthenia | 98 | 80 | 71

18. Secondary Outcome: STAGE-I: Number of Participants With Solicited Systemic Reactions Following Vaccination With CYD Dengue Vaccine or Placebo (Post Each Vaccination)
Description: An AR was defined as all noxious and unintended responses to a medicinal product related to any dose. A SR was defined as an AR observed and reported under the conditions (symptom and onset) prelisted (i.e., solicited) in the eCRF and considered as related to vaccination. Solicited systemic reactions included fever, headache, malaise, myalgia, and asthenia.
Time Frame: Within 14 days after each vaccination (1, 2, and 3)
Population: Analysis was performed on SafAS. Here, 'Number analyzed'=participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | STAGE-I Group 1: CYD Dengue Vaccine | STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12) | STAGE-I Group 3: Placebo + CYD Dengue Vaccine (Month 12)
Number analyzed (Participants) | 347 | 347 | 352
Participants
  Post-vaccination 1: Fever | 10 | 8 | 13
  Post-vaccination 1: Headache | 90 | 83 | 84
  Post-vaccination 1: Malaise | 74 | 60 | 61
  Post-vaccination 1: Myalgia | 67 | 55 | 48
  Post-vaccination 1: Asthenia | 63 | 52 | 45
  Post-vaccination 2: Fever: number analyzed (Participants) | 332 | 327 | 330
  Post-vaccination 2: Fever | 12 | 7 | 12
  Post-vaccination 2: Headache: number analyzed (Participants) | 332 | 328 | 332
  Post-vaccination 2: Headache | 54 | 55 | 53
  Post-vaccination 2: Malaise: number analyzed (Participants) | 332 | 328 | 332
  Post-vaccination 2: Malaise | 50 | 44 | 47
  Post-vaccination 2: Myalgia: number analyzed (Participants) | 332 | 328 | 332
  Post-vaccination 2: Myalgia | 49 | 33 | 35
  Post-vaccination 2: Asthenia: number analyzed (Participants) | 332 | 328 | 332
  Post-vaccination 2: Asthenia | 40 | 30 | 33
  Post-vaccination 3: Fever: number analyzed (Participants) | 324 | 317 | 317
  Post-vaccination 3: Fever | 9 | 8 | 9
  Post-vaccination 3: Headache: number analyzed (Participants) | 325 | 321 | 324
  Post-vaccination 3: Headache | 55 | 47 | 47
  Post-vaccination 3: Malaise: number analyzed (Participants) | 325 | 321 | 324
  Post-vaccination 3: Malaise | 46 | 41 | 39
  Post-vaccination 3: Myalgia: number analyzed (Participants) | 325 | 321 | 324
  Post-vaccination 3: Myalgia | 26 | 37 | 28
  Post-vaccination 3: Asthenia: number analyzed (Participants) | 325 | 321 | 324
  Post-vaccination 3: Asthenia | 29 | 32 | 21

19. Secondary Outcome: STAGE-II: Number of Participants With Solicited Injection Site Reactions Following Booster Vaccination With CYD Dengue Vaccine
Description: An AR was defined as all noxious and unintended responses to a medicinal product related to any dose. A SR was defined as an AR observed and reported under the conditions (symptom and onset) prelisted (i.e., solicited) in the eCRF and considered as related to vaccination. Solicited injection site reaction was an AR at and around the injection site that included pain, erythema, and swelling.
Time Frame: Within 7 days after CYD booster vaccination
Population: Analysis was performed on SafAS. Here, 'Number analyzed'=participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | STAGE-II Group 1a: CYD Vaccine + CYD Booster Vaccine (1 Year) | STAGE-II Group 2a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 3a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 1b: CYD Vaccine + CYD Booster Vaccine (2 Years) | STAGE-II Group 2b: Placebo + CYD + CYD Booster (2 Years) | STAGE-II Group 3b: Placebo + CYD + CYD Booster (2 Years)
Number analyzed (Participants) | 55 | 59 | 62 | 53 | 54 | 52
Participants
  Pain | 6 | 7 | 11 | 7 | 12 | 10
  Erythema | 0 | 0 | 0 | 0 | 1 | 0
  Swelling | 0 | 0 | 0 | 0 | 1 | 1

20. Secondary Outcome: STAGE-II: Number of Participants With Solicited Systemic Reactions Following Booster Vaccination With CYD Dengue Vaccine
Description: as for outcome 18
Time Frame: Within 14 days after CYD booster vaccination
Population: Analysis was performed on SafAS. Here, 'Number analyzed'=participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | STAGE-II Group 1a: CYD Vaccine + CYD Booster Vaccine (1 Year) | STAGE-II Group 2a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 3a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 1b: CYD Vaccine + CYD Booster Vaccine (2 Years) | STAGE-II Group 2b: Placebo + CYD + CYD Booster (2 Years) | STAGE-II Group 3b: Placebo + CYD + CYD Booster (2 Years)
Number analyzed (Participants) | 55 | 59 | 62 | 53 | 54 | 52
Participants
  Fever: number analyzed (Participants) | 55 | 59 | 62 | 53 | 54 | 51
  Fever | 1 | 0 | 1 | 2 | 2 | 0
  Headache | 5 | 11 | 6 | 7 | 11 | 7
  Malaise | 5 | 9 | 7 | 7 | 9 | 5
  Myalgia | 5 | 8 | 9 | 9 | 12 | 6
  Asthenia | 4 | 6 | 6 | 7 | 9 | 3

21. Secondary Outcome: STAGE-I: Number of Participants Reporting Unsolicited Adverse Events Following Vaccination With CYD Dengue Vaccine or Placebo
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the eCRF in terms of diagnosis and/or onset post-vaccination.
Time Frame: Within 28 days after any vaccination (1, 2, or 3)
Population: Analysis was performed on SafAS.
Measure: Count of Participants; unit: Participants
Arm/Group | STAGE-I Group 1: CYD Dengue Vaccine | STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12) | STAGE-I Group 3: Placebo + CYD Dengue Vaccine (Month 12)
Number analyzed (Participants) | 348 | 348 | 352
Participants | 73 | 94 | 75

22. Secondary Outcome: STAGE-II: Number of Participants Reporting Unsolicited Adverse Events Following Booster Vaccination With CYD Dengue Vaccine
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An unsolicited AE was an observed AE that does not fulfill the conditions prelisted in the eCRF in terms of diagnosis and/or onset post-vaccination.
Time Frame: Within 28 days after CYD booster Vaccination
Population: Analysis was performed on SafAS.
Measure: Count of Participants; unit: Participants
Arm/Group | STAGE-II Group 1a: CYD Vaccine + CYD Booster Vaccine (1 Year) | STAGE-II Group 2a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 3a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 1b: CYD Vaccine + CYD Booster Vaccine (2 Years) | STAGE-II Group 2b: Placebo + CYD + CYD Booster (2 Years) | STAGE-II Group 3b: Placebo + CYD + CYD Booster (2 Years)
Number analyzed (Participants) | 55 | 59 | 62 | 53 | 56 | 53
Participants | 1 | 3 | 5 | 3 | 2 | 4

23. Secondary Outcome: STAGE-I: Number of Participants Reporting Serious Adverse Events Including Serious Adverse Event of Special Interests (AESI) Following Vaccination With CYD Dengue Vaccine or Placebo
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was congenital anomaly/birth defect, or was an important medical event. AESI were AEs that were considered by the Sponsor to be relevant for the monitoring of the safety profile of the investigational vaccine.
Time Frame: From Day 0 (post vaccination) up to 12 months after last vaccination in STAGE-I (i.e., up to 24 months)
Population: Analysis was performed on SafAS.
Measure: Count of Participants; unit: Participants
Arm/Group | STAGE-I Group 1: CYD Dengue Vaccine | STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12) | STAGE-I Group 3: Placebo + CYD Dengue Vaccine (Month 12)
Number analyzed (Participants) | 348 | 348 | 352
Participants
  SAE | 14 | 26 | 18
  Serious AESI | 0 | 0 | 0

24. Secondary Outcome: STAGE-II: Number of Participants Reporting Serious Adverse Events Including Serious Adverse Events Special Interest Following Booster Vaccination With CYD Dengue Vaccine
Description: as for outcome 23
Time Frame: From Month 25 up to 6 months after CYD booster injection (either at 1 year or 2 year) (i.e., up to 30 months for Groups 1a, 2a, and 3a and up to 42 months for Groups 1b, 2b, and 3b)
Population: Analysis was performed on SafAS.
Measure: Count of Participants; unit: Participants
Arm/Group | STAGE-II Group 1a: CYD Vaccine + CYD Booster Vaccine (1 Year) | STAGE-II Group 2a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 3a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 1b: CYD Vaccine + CYD Booster Vaccine (2 Years) | STAGE-II Group 2b: Placebo + CYD + CYD Booster (2 Years) | STAGE-II Group 3b: Placebo + CYD + CYD Booster (2 Years)
Number analyzed (Participants) | 55 | 59 | 62 | 53 | 56 | 53
Participants
  SAE | 3 | 0 | 2 | 2 | 0 | 1
  Serious AESI | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Unsolicited non-serious AEs: Day 0 to Day 28 post any vaccination SR: within 7 & 14 days post any vaccination; SAE: up to 24 months for STAGE-I); up to 6 months after last vaccination for Stage-2 (i.e., up to 30 months [for Groups 1a, 2a, and 3a]; & up to 42 months [for Groups 1b, 2b, and 3b])
Description: Analysis was performed on SafAS. SR was AE that was prelisted (i.e., solicited) in the eCRF and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e., solicited) in the eCRF in terms of symptom and/or onset post-vaccination. Reported AEs were presented as pre-specified in the study protocol.
Groups:
- STAGE-II Group 1a: CYD Vaccine + CYD Booster Vaccine (1 Year): Participants from Group 1 who received vaccination in STAGE-I and were seropositive at Baseline received a booster dose of CYD dengue vaccine in STAGE-II at 1 year post last dose in STAGE-I (i.e. at Month 24).
- STAGE-II Group 1b: CYD Vaccine + CYD Booster Vaccine (2 Years): Participants from Group 1 who received vaccination in STAGE-I and were seropositive at baseline received a booster injection of CYD dengue vaccine in STAGE-II at 2 years post last dose in STAGE-I (i.e. at Month 36).
- STAGE-II Group 2a: Placebo + CYD + CYD Booster (1 Year): Participants from Group 2 who received vaccination in STAGE-I and were seropositive at baseline received a booster injection of CYD dengue vaccine in STAGE-II at 1 year post last dose in STAGE-I (i.e. at Month 24).
- STAGE-II Group 2b: Placebo + CYD + CYD Booster (2 Years): Participants from Group 2 who received vaccination in STAGE-I and were seropositive at baseline received a booster injection of CYD dengue vaccine in STAGE-II at 2 years post last dose in STAGE-I (i.e. at Month 36).
- STAGE-II Group 3a: Placebo + CYD + CYD Booster (1 Year): Participants from Group 3 who received vaccination in STAGE-I and were seropositive at baseline received a booster injection of CYD dengue vaccine in STAGE-II at 1 year post last dose in STAGE-I (i.e. at Month 24).
- STAGE-II Group 3b: Placebo + CYD + CYD Booster (2 Years): Participants from Group 3 who received vaccination in STAGE-I and were seropositive at baseline received a booster injection of CYD dengue vaccine in STAGE-II at 2 years post last dose in STAGE-I (i.e. at Month 36).
Arm/Group | STAGE-I Group 1: CYD Dengue Vaccine | STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12) | STAGE-I Group 3: Placebo + CYD Dengue Vaccine (Month 12) | STAGE-II Group 1a: CYD Vaccine + CYD Booster Vaccine (1 Year) | STAGE-II Group 1b: CYD Vaccine + CYD Booster Vaccine (2 Years) | STAGE-II Group 2a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 2b: Placebo + CYD + CYD Booster (2 Years) | STAGE-II Group 3a: Placebo + CYD + CYD Booster (1 Year) | STAGE-II Group 3b: Placebo + CYD + CYD Booster (2 Years)
All-Cause Mortality (participants affected / at risk) | 0/348 | 1/348 | 1/352 | 0/55 | 0/53 | 0/59 | 0/56 | 0/62 | 0/53
Serious Adverse Events (participants affected / at risk) | 14/348 | 26/348 | 18/352 | 3/55 | 2/53 | 0/59 | 0/56 | 2/62 | 1/53
Other Adverse Events (participants affected / at risk) | 203/348 | 189/348 | 182/352 | 10/55 | 13/53 | 15/59 | 20/56 | 18/62 | 15/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STAGE-I Group 1: CYD Dengue Vaccine (N=348) | STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12) (N=348) | STAGE-I Group 3: Placebo + CYD Dengue Vaccine (Month 12) (N=352) | STAGE-II Group 1a: CYD Vaccine + CYD Booster Vaccine (1 Year) (N=55) | STAGE-II Group 1b: CYD Vaccine + CYD Booster Vaccine (2 Years) (N=53) | STAGE-II Group 2a: Placebo + CYD + CYD Booster (1 Year) (N=59) | STAGE-II Group 2b: Placebo + CYD + CYD Booster (2 Years) (N=56) | STAGE-II Group 3a: Placebo + CYD + CYD Booster (1 Year) (N=62) | STAGE-II Group 3b: Placebo + CYD + CYD Booster (2 Years) (N=53)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Branchial Cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid Cyst (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea Infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis A (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Animal Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Forearm Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gun Shot Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaw Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid Haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion Spontaneous Incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Threatened Labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus Urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal Colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bartholin's Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine Polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic Skin Eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STAGE-I Group 1: CYD Dengue Vaccine (N=348) | STAGE-I Group 2: Placebo + CYD Dengue Vaccine (Months 6,12) (N=348) | STAGE-I Group 3: Placebo + CYD Dengue Vaccine (Month 12) (N=352) | STAGE-II Group 1a: CYD Vaccine + CYD Booster Vaccine (1 Year) (N=55) | STAGE-II Group 1b: CYD Vaccine + CYD Booster Vaccine (2 Years) (N=53) | STAGE-II Group 2a: Placebo + CYD + CYD Booster (1 Year) (N=59) | STAGE-II Group 2b: Placebo + CYD + CYD Booster (2 Years) (N=56) | STAGE-II Group 3a: Placebo + CYD + CYD Booster (1 Year) (N=62) | STAGE-II Group 3b: Placebo + CYD + CYD Booster (2 Years) (N=53)
Asthenia (General disorders) | 98 (133) | 80 (114) | 71 (100) | 4 (4) | 7 (7) | 6 (6) | 9 (9) | 6 (6) | 3 (3)
Fever (General disorders) | 29 (31) | 21 (23) | 31 (34) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Injection Site Pain (General disorders) | 109 (154) | 114 (164) | 97 (146) | 6 (6) | 7 (7) | 7 (7) | 12 (12) | 11 (11) | 10 (10)
Malaise (General disorders) | 114 (170) | 98 (146) | 103 (148) | 5 (5) | 7 (7) | 9 (9) | 9 (9) | 7 (7) | 5 (5) — Events of malaise that occurred after 14 days post-vaccination were considered as unsolicited AE.
Myalgia (Musculoskeletal and connective tissue disorders) | 110 (143) | 92 (126) | 87 (112) | 5 (5) | 9 (9) | 8 (8) | 12 (12) | 9 (9) | 6 (6) — Events of myalgia that occurred after 14 days post-vaccination were considered as unsolicited AE.
Headache (Nervous system disorders) | 129 (201) | 123 (190) | 124 (184) | 5 (5) | 7 (7) | 11 (11) | 12 (12) | 7 (7) | 7 (7) — Events of headache that occurred after 14 days post-vaccination were considered as unsolicited AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT02628444/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT02628444/SAP_001.pdf